CLINICAL TRIAL: NCT00495326
Title: Randomized Non-inferiority Trial Comparing the Nevirapine-based Antiretroviral Therapy Versus the Standard Efavirenz-based ART for the Treatment of HIV-TB Co-infected Patients on Rifampicin-based Therapy (ANRS 12146 CARINEMO)
Brief Title: Comparison of Nevirapine and Efavirenz for the Treatment of HIV-TB Co-infected Patients (ANRS 12146 CARINEMO)
Acronym: CARINEMO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12146 CARINEMO
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Tuberculosis; Aids; Hiv Infections
Keywords: drug interactions; Treatment Naive
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — stavudine, lamivudine, nevirapine drug combination; Rifampin; Ethambutol; Isoniazid; Protons; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Nevirapine-based ART
  Interventions: Drug: Nevirapine based therapy; Drug: Rifampicin (RMP) Ethambutol (E) Isoniazid (H) Pyrazinamid (Z)
- 2 (Active Comparator): Efavirenz-based ART
  Interventions: Drug: Efavirenz based therapy; Drug: Rifampicin (RMP) Ethambutol (E) Isoniazid (H) Pyrazinamid (Z)

INTERVENTIONS:
Drug: Nevirapine based therapy — * Patients below 60 kg: 1 tablet twice a day of Triomune30®, including NVP 200 mg, 3TC 150 mg and D4T 30mg
  * Patients above 60kg: 1 tablet twice a day of Triomune40®, including NVP 200 mg, 3TC 150 mg and D4T 40 mg)
  Other Names: Triomune
  Arms: 1
Drug: Efavirenz based therapy — Efavirenz EFV 200 mg (3 tablets/d) Lamivudine 3TC 300mg (2 tablets of 150mg/d) D4T generic 30mg or 40mg (2 tablets/d)
  Other Names: Stockrin; Cipla drugs
  Arms: 2
Drug: Rifampicin (RMP) Ethambutol (E) Isoniazid (H) Pyrazinamid (Z) — * Intensive phase: 2 months daily E(RMP)HZ. PTB smear positive patients at month 2 will receive 1 more month intensive phase.
  * Continuation phase: 4 months daily H(RMP).
  * Patients with meningitis will receive Streptomycin instead of E during intensive phase.

SUMMARY:
The purpose of this study is to determine whether the use of Nevirapine in HIV patients already treated against tuberculosis by Rifampicin is as efficient and as well tolerated as Efavirenz.

DETAILED DESCRIPTION:
Anti Retroviral Therapy (ART) reduces tuberculosis (TB) incidence in HIV-infected patients and reduces mortality among TB patients with deep immune suppression. The Fixed Drug Combination (FDC) nevirapine (NVP)-lamivudine-stavudine is the first line ART available for low-income countries. Rifampicin (RMP), due to its liver induction effect, reduces significantly NVP plasma concentration, raising concerns regarding the risk of resistance and subsequent treatment failure. Therefore, in co-infected patients, WHO recommends delaying ART or using efavirenz (EFV)-based ART. Although EFV is also reduced at lower level, longitudinal studies report good efficacy and safety when given concomitantly with RMP.

In low-income countries, poor access to EFV, contradiction during pregnancy and absence of FDC containing EFV lead to difficulties in HIV-TB treatment.

Despite 2 limited retrospective studies and a non-randomised prospective study, which report good virological response at 6 months in co-infected patients receiving NVP and RMP co-administration, existing data are too limited to change the recommendation.

The aim of the study is to compare, in terms of therapeutic efficacy and clinical safety, the nevirapine-based HAART to the standard efavirenz-based HAART, in HIV/TB co-infected patients receiving a rifampicin-based TB treatment.

The study will evaluate one year after TB treatment initiation, whether the HAART efficacy (virological outcome, death or lost of follow-up) induced by NVP-based HAART is non-inferior to those induced by EFV based HAART, in patients receiving concomitantly HAART and RMP-based TB treatment.

ELIGIBILITY:
Inclusion Criteria:

* Person HIV infected
* Aged of 18 years or more
* Signed informed consent
* New case of tuberculosis: patient who never received TB treatment or for less than 1 month
* Patients receiving rifampicin based TB regimen since 4 to 6 weeks
* CD4 cell count < 250 cell/mm3 in the 4 weeks following the TB diagnosis
* Naïve of HAART
* For women of childbearing age, to have a negative plasmatic test for pregnancy and to accept to take a contraception or declare no wish of pregnancy in the coming year.

Exclusion Criteria:

* To have a positive plasmatic test for pregnancy
* Karnofsky score <60%
* ALAT > 4N (Hepatitis grade 3 or 4)
* Ongoing psychiatric pathology
* Refuse to participate in the study

Amendment :

* bilirubin > grade 3
* any grade 4 clinical sign or biological result at time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2007-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Viral load measure (Virological failure will be defined after 2 consecutive measures as : More than 1 log10 increase in plasma HIV-1 RNA concentration for patients with detectable viral load (> 50 copies/mL) at the previous dosage.) | 3, 6 and 12 months

SECONDARY OUTCOMES:
New or recurrent stage 3 or 4 HIV/AIDS related events | 12 months
Deaths after one year | 12 months
Severe drugs side effects | 12 months
Immune Reconstitution Syndrome(IRIS) | 12 months
Increase of CD4 cell count induced by HAART | at 6 months and 1 year
Pharmacokinetic profile of nevirapine when combined with rifampicin | 2 months
Rifampicin plasma concentration dosage | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Maryline Bonnet, MD, Principal Investigator — Epicentre; Nilesh Bhatt, MD, Principal Investigator — Ministry of Health, Instituto Nacional de Saude, Mozambique
Locations (3):
- Mozambique (3):
  - Health centre of Alto Mae, Chamanculo district, Maputo
  - Health centre of Josue Macao, Maputo
  - Health centre of Malavane, Maputo

REFERENCES:
- [Derived] Bhatt NB, Barau C, Amin A, Baudin E, Meggi B, Silva C, Furlan V, Grinsztejn B, Barrail-Tran A, Bonnet M, Taburet AM; ANRS 12146-CARINEMO Study Group. Pharmacokinetics of rifampin and isoniazid in tuberculosis-HIV-coinfected patients receiving nevirapine- or efavirenz-based antiretroviral treatment. Antimicrob Agents Chemother. 2014 Jun;58(6):3182-90. doi: 10.1128/AAC.02379-13. Epub 2014 Mar 24. PMID 24663014
- [Derived] Bonnet M, Bhatt N, Baudin E, Silva C, Michon C, Taburet AM, Ciaffi L, Sobry A, Bastos R, Nunes E, Rouzioux C, Jani I, Calmy A; CARINEMO study group. Nevirapine versus efavirenz for patients co-infected with HIV and tuberculosis: a randomised non-inferiority trial. Lancet Infect Dis. 2013 Apr;13(4):303-12. doi: 10.1016/S1473-3099(13)70007-0. Epub 2013 Feb 20. PMID 23433590
- See also: Related Info — http://www.anrs.fr